CLINICAL TRIAL: NCT00965848
Title: A Post Marketing Surveillance Study on the Safety and Effectiveness of Doripenem in the Therapy of Thai Patients With Nosocomial Pneumonia, Complicated Intra-Abdominal Infections and Complicated Urinary Tract Infections
Brief Title: A Safety and Efficacy Study of Doripenem in Participants With Nosocomial Pneumonia, Complicated Intra-Abdominal Infections and Urinary Tract Infections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen-Cilag Ltd.,Thailand (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR015766; DORIBAC4003
Record Dates: First submitted 2009-08-24; First posted 2009-08-26 (Estimated); Results first posted 2013-08-28 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-09

CONDITIONS: Infection; Cross Infection; Bacterial Infections; Pneumonia, Ventilator-Associated; Intra-abdominal Infections; Urinary Tract Infections
Keywords: Pneumonia, Ventilator-Associated; Intra-abdominal Infections; Urinary tract Infections; Doripenem; Doribax
MeSH Terms: conditions — Infections; Cross Infection; Bacterial Infections; Pneumonia, Ventilator-Associated; Intraabdominal Infections; Urinary Tract Infections | interventions — Doripenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nosocomial Pneumonia (Experimental): Doripenem will be administered as 1 or 4 hours intravenous infusion at a dose of 500 mg every 8 hours in participants with nosocomial pneumonia up to maximum of 14 days.
  Interventions: Drug: Doripenem
- Complicated Intra-Abdominal Infections (Experimental): Doripenem will be administered as 1 or 4 hours intravenous infusion at a dose of 500 mg every 8 hours in participants with complicated intra-abdominal infections up to maximum of 14 days.
  Interventions: Drug: Doripenem
- Complicated Urinary Tract Infections (Experimental): Doripenem will be administered as 1 or 4 hours intravenous infusion at a dose of 500 mg every 8 hours in participants with complicated urinary tract infections up to maximum of 10 days.
  Interventions: Drug: Doripenem

INTERVENTIONS:
Drug: Doripenem — Doripenem 500 mg will be administered as 1 or 4 hours intravenous infusion, after every 8 hours up to maximum of 14 days.
  Other Names: Doribax

SUMMARY:
The purpose of this study is to assess the safety and efficacy of doripenem in participants with nosocomial pneumonia (inflammation of the lungs in which the lungs become heavy; pneumonia occurring at least 48 hours after hospital admission), complicated intra-abdominal (in belly) infections and complicated urinary tract infections (bladder infections).

DETAILED DESCRIPTION:
This is an open-label (all people involved know the identity of the intervention), multi-center (conducted in more than 1 center) study, to evaluate the safety and effectiveness of doripenem in treating Thai participants with nosocomial pneumonia, complicated intra-abdominal and urinary tract infections. The study consists of 4 visits: Visit 1 (Baseline), Visit 2 (End-of-Treatment [EOT], up to Day 14), Visit 3 (Phone visit, Test-of-Cure [TOC], up to Day 14 after EOT) and Visit 4 (Phone visit, Day 90). Participants will receive 500 milligram (mg) of doripenem as intravenous infusion (directly into the vein) every 8 hours for at least 3 days after clinical response and extended up to 14 days. Efficacy will primarily be evaluated by determination of clinical response. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Eligibility Criteria:

Inclusion Criteria:

* Male or female participants with 18 years old age and above
* Diagnosed nosocomial pneumonia, complicated intra-abdominal infections and complicated urinary tract infections
* Must have evidence of a systemic inflammatory response syndrome with at least one of the these: fever (body temperature greater than 38 degree celcius) or hypothermia (body temperature less than 36 degree celcius) or elevated total peripheral white blood cell count greater than or equal to 12,000 cells per cubic millimeter or leukopenia with less than 4,000 cells per cubic millimeter or decrease in blood pressure relative to Baseline of greater than 15 millimeter of mercury systolic or increased pulse greater than 100 beats per minute (bpm) and respiratory rates greater than 20 bpm
* Candidate for treatment with carbapenems, with at least one of these conditions: Empirical therapy; suspected infection caused by carbapenem susceptible P. aeruginosa or carbapenem-susceptible A. baumannii or MDR gram negative bacteria or nosocomial infection with failure of previous treatment or modified therapy; known pathogens with resistance to cephalosporins,aminoglycosides, fluoroquinolones or beta-lactam/ batalactamase intibitor and susceptible to carbapenem or known infection caused by gram negative bacteria
* Signed informed consent

Exclusion Criteria:

* Pregnant or lactating female participants
* History of severe allergies to antibiotics such as penicillins, cephalosporins and carbapenems
* Hypersensitivity to doripenem and/or excipients
* Previous use of carbapenems within 7 days of study entry
* Participants in terminal stage of malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2009-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Ltd.,Thailand Clinical Trial, Study Director — Janssen-Cilag Ltd.,Thailand
Locations (8):
- Thailand (8):
  - Bangkok
  - Chiang Mai
  - Chiang Rai
  - Chon Buri
  - Khon Kaen
  - Nakhon Ratchasima
  - Nakornnayok
  - Pathum Thani

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The total number of participants enrolled were 270, out of which 268 participants had adequate information for analysis.
Groups:
- Nosocomial Pneumonia: Doripenem was administered as 1 or 4 hours intravenous infusion (directly into the vein) at a dose of 500 milligram (mg) every 8 hours in participants with nosocomial pneumonia up to maximum of 14 days.
- Complicated Intra-Abdominal Infections: Doripenem was administered as 1 or 4 hours intravenous infusion at a dose of 500 mg every 8 hours in participants with complicated intra-abdominal infections up to maximum of 14 days.
- Complicated Urinary Tract Infections: Doripenem was administered as 1 or 4 hours intravenous infusion at a dose of 500 mg every 8 hours in participants with complicated urinary tract infections up to maximum of 10 days.
Period: Overall Study
Arm/Group | Nosocomial Pneumonia | Complicated Intra-Abdominal Infections | Complicated Urinary Tract Infections
Started | 107 | 34 | 127
Completed | 78 | 32 | 117
Not Completed | 29 | 2 | 10
Not completed — Protocol Violation | 3 | 0 | 1
Not completed — Death | 11 | 1 | 5
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Indeterminate Clinical Outcome | 2 | 0 | 1
Not completed — Not Clinically Evaluable | 7 | 1 | 1
Not completed — Other | 5 | 0 | 1

BASELINE CHARACTERISTICS:
Population: For Baseline characteristics, age and gender, number of participants evaluable was 264.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 264
Age Continuous [Mean (Standard Deviation); unit: Years] | 64.6 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118
  Male | 146

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Number of Participants Discontinued Because of AEs
Description: An adverse event is any untoward medical occurrence in a participant administered with a pharmaceutical product. An adverse event does not necessarily have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. The number of participants discontinued because of AEs were also reported.
Time Frame: Up to 30 days after last dose of study drug
Population: Intent-to-treat population (ITT) included all participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Nosocomial Pneumonia | Complicated Intra-Abdominal Infections | Complicated Urinary Tract Infections
Number analyzed (Participants) | 107 | 34 | 127
Participants
  Participants with AEs | 66 | 22 | 56
  Participants discontinued because of AEs | 0 | 0 | 2

2. Secondary Outcome: Percentage of Participants With Clinical Response at End-of-Treatment (EOT)
Description: Clinical response was defined as cure, improvement, failure and indeterminate. Cure=All signs/symptoms resolved/improved/lack of progression of all abnormalities; Improvement=Signs/symptoms of disease improved/resolved/ no modification in antibiotic therapy required & no worsening/appearance of new signs & symptoms of disease; Failure=Persistence or worsening of signs/symptoms of disease or emergence of new signs/symptoms and require any other antimicrobial therapy; and Indeterminate=Insufficient data for treatment evaluation. 2 subjects were lost to follow-up.
Time Frame: Up to Day 14 (EOT)
Population: Clinical Modified-Intent-to-Treat (cMITT) included all participants who received any dose of study medication. "N" signifies those participants who were evaluated for this measure at the specified time point for each arm group respectively.
Measure: Number; unit: Percentage of participants
Arm/Group | Nosocomial Pneumonia | Complicated Intra-Abdominal Infections | Complicated Urinary Tract Infections
Number analyzed (Participants) | 97 | 33 | 125
Percentage of participants
  Cure | 38.1 | 57.6 | 71.2
  Improvement | 30.9 | 33.3 | 20.8
  Failure | 11.3 | 6.1 | 1.6
  Indeterminate | 18.6 | 3.0 | 5.6
  Other: Lost to Follow-Up | 1.0 | 0.0 | 0.8

3. Secondary Outcome: Percentage of Participants With Clinical Response at Test-of-Cure (TOC)
Description: Clinical response was defined as cure, improvement, failure and indeterminate. Cure=All signs/symptoms resolved/improved/lack of progression of all abnormalities; Improvement=Signs/symptoms of disease improved/resolved/ no modification in antibiotic therapy required and no worsening/appearance of new signs & symptoms of disease; Failure=Persistence or worsening of signs/symptoms of disease or emergence of new signs/symptoms & require any other antimicrobial therapy; & Indeterminate=Insufficient data for treatment evaluation. The TOC visit (up to Day 14 after EOT) was conducted by phone. Participants who were assessed as cure or improvement at EOT will be evaluated for clinical response at TOC (up to Day 14 after EOT).
Time Frame: Up to Day 14 after End-of-Treatment (EOT)
Population: The cMITT included all participants who received any dose of study medication. "N" signifies those participants who were evaluated for this measure at the specified time point for each arm group respectively.
Measure: Number; unit: Percentage of Participants
Arm/Group | Nosocomial Pneumonia | Complicated Intra-Abdominal Infections | Complicated Urinary Tract Infections
Number analyzed (Participants) | 62 | 24 | 93
Percentage of Participants
  Cure | 56.96 | 66.67 | 85.42
  Improvement | 0.00 | 0.00 | 0.00
  Failure | 5.06 | 7.41 | 6.25
  Indeterminate | 15.19 | 14.81 | 5.21
  Other: Lost to Follow-Up | 1.27 | 0.00 | 0.00
  Not evaluable | 21.52 | 11.11 | 3.13

4. Secondary Outcome: Number of Participants With 90-day Mortality
Description: Number of Participants with 90-day mortality was defined as the number of participants who died by Day 90.
Time Frame: up to Day 90
Population: The cMITT included all participants who received any dose of study medication and met the clinical definition in the protocol. "N" signifies those participants who were evaluated for this measure.
Measure: Number; unit: Participants
Arm/Group | Nosocomial Pneumonia | Complicated Intra-Abdominal Infections | Complicated Urinary Tract Infections
Number analyzed (Participants) | 89 | 34 | 116
Participants | 42 | 16 | 22

ADVERSE EVENTS:
Time Frame: Baseline up to 30 days after last dose of study drug
Description: An adverse event is any untoward medical occurrence in a clinical study participant administered with study treatment. It can be any unfavorable and unintended sign/abnormal finding, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Arm/Group | Nosocomial Pneumonia | Complicated Intra-Abdominal Infections | Complicated Urinary Tract Infections
Serious Adverse Events (participants affected / at risk) | 45/107 | 14/34 | 31/127
Other Adverse Events (participants affected / at risk) | 66/107 | 22/34 | 56/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nosocomial Pneumonia (N=107) | Complicated Intra-Abdominal Infections (N=34) | Complicated Urinary Tract Infections (N=127)
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Right ventricular failure (Cardiac disorders) | 1 | 0 | 0
Sudden cardiac death (Cardiac disorders) | 3 | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 3 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1 | 2
Colorectal cancer (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1 | 0
Pancreatic carcinoma (Gastrointestinal disorders) | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1
Peritonitis (Gastrointestinal disorders) | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 1
Multi-organ failure (General disorders) | 0 | 4 | 0
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0
Bile duct cancer (Hepatobiliary disorders) | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic neoplasm malignant (Hepatobiliary disorders) | 0 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1
Acquired immunodeficiency syndrome (Infections and infestations) | 1 | 0 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0 | 0
Catheter related infection (Infections and infestations) | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1
Fungal sepsis (Infections and infestations) | 0 | 0 | 1
HIV infection (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 10 | 2 | 4
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 7 | 5 | 3
Septic shock (Infections and infestations) | 10 | 4 | 9
Urinary tract infection (Infections and infestations) | 1 | 0 | 3
Urosepsis (Infections and infestations) | 0 | 0 | 1
Wound infection (Infections and infestations) | 1 | 0 | 0
Wound sepsis (Infections and infestations) | 0 | 1 | 0
Drug prescribing error (Injury, poisoning and procedural complications) | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Myasthenias (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1
Bladder cancer (Renal and urinary disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 2 | 1 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung cancer metastatic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung neoplasm malignant (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 2 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nosocomial Pneumonia (N=107) | Complicated Intra-Abdominal Infections (N=34) | Complicated Urinary Tract Infections (N=127)
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 1 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 2
Ileus (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 2
Oral candidiasis (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 3
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic encephalopathy (Hepatobiliary disorders) | 0 | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0 | 0
Drug eruption (Immune system disorders) | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0
Abdominal infection (Infections and infestations) | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1
Candida sepsis (Infections and infestations) | 0 | 0 | 1
Catheter related infection (Infections and infestations) | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0
Fungal cystitis (Infections and infestations) | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 2 | 3
Sepsis (Infections and infestations) | 0 | 0 | 1
Septic shock (Infections and infestations) | 1 | 0 | 0
Skin candida (Infections and infestations) | 0 | 0 | 1
Skin infection (Infections and infestations) | 2 | 0 | 1
Stenotrophomonas infection (Infections and infestations) | 1 | 0 | 0
Strongyloidiasis (Infections and infestations) | 1 | 0 | 0
Systemic candida (Infections and infestations) | 0 | 0 | 1
Tinea cruris (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 4
Urinary tract infection enterococcal (Infections and infestations) | 0 | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 1
Application site itching (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 2 | 0 | 0
Blood urea increased (Investigations) | 1 | 1 | 1
Hepatic enzyme increased (Investigations) | 3 | 1 | 1
Transaminase increased (Investigations) | 1 | 0 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 2 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypothyroidism (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Gout (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Convulsion (Nervous system disorders) | 2 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 2
Insomnia (Nervous system disorders) | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Pyuria (Renal and urinary disorders) | 0 | 0 | 2
Renal failure acute (Renal and urinary disorders) | 4 | 0 | 2
Urinary tract infection (Renal and urinary disorders) | 1 | 0 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Tracheobronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Cellulitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 5 | 1 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Tracheostomy (Surgical and medical procedures) | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1
Phlebitis (Vascular disorders) | 2 | 2 | 1
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If the Institution & Principal Investigator wish to publish information from Clinical Trial, a copy of manuscript must be provided to Sponsor at least 60 days prior to submission for publication/presentation & will arrange expedited reviews for the same. No paper with confidential Information will be submitted without Sponsor's prior consent. If requested, Institution & Principal Investigator will hold such publication for up to additional 60 days to allow filing of patent application.